CLINICAL TRIAL: NCT05978362
Title: Prospective, Multicenter, Randomized Single-blind Study on the Interest of Capsular Repair in the Latarjet Operation
Brief Title: Value of Capsular Repair for Latarjet
Acronym: CAP-LATARJET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A02629-34
Record Dates: First submitted 2023-07-18; First posted 2023-08-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: prospective, comparative, longitudinal, randomized single-blind study
Who Masked: Participant
Masking Description: randomized single-blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With capsular repair (Experimental): This technique consists of inserting the capsule during the operation according to Latarjet.
  Interventions: Procedure: Latarjet technique
- Without capsular repair (Active Comparator): Latarjet technique without capsular repair
  Interventions: Procedure: Latarjet technique

INTERVENTIONS:
Procedure: Latarjet technique — Realization of a stop according to Latarjet

SUMMARY:
The purpose of the study is to evaluate the occurrence of osteoarthritis (YES/NO) by radiography.

DETAILED DESCRIPTION:
This is a prospective, comparative, longitudinal, randomized, single-blind, multicenter study.

This study will validate preliminary results on a technique associating capsular repair with abutment according to Latarjet in the treatment of shoulder instabilities. It may help reduce the risk of osteoarthritis and thus allow patients to maintain a healthy, stable and painless shoulder for longer.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over the age of 18
* Patient with shoulder instability with risk factors for recurrence (ISIS score > 3), requiring surgical stabilization by abutment
* Affiliated patient or beneficiary of a social security scheme
* Patient having been informed and having given his free, informed and written consent.

Exclusion Criteria:

* Patient with history of surgery for instability of the same shoulder
* Patient presenting contraindications to the realization of a postoperative scanner
* Patient whose physical and/or psychological health is severely impaired, which according to the investigator may affect the compliance of the study participant
* Patient participating in another clinical research or in a period of exclusion from another research still in progress at the time of inclusion
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of osteoarthritis | 10 years
  Change from occurrence of osteoarthritis (YES/NO) on X-ray at 5 and 10 years, compared to inclusion X-ray using the Samilson-Prieto classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Maussins-Nollet, Paris, France